CLINICAL TRIAL: NCT06145789
Title: The Use of Standing Powered Wheelchairs in Individuals With Spinal Cord Injury
Brief Title: The Use of Standing Powered Wheelchairs in Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Örücü Atar, Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E1-23-4267
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries
Keywords: standing powered wheelchair; spinal cord injury; satisfaction; secondary complication
MeSH Terms: conditions — Spinal Cord Injuries; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- standing powered wheelchair: standing powered wheelchair evaluation
  Interventions: Other: standing powered wheelchair evaluation

INTERVENTIONS:
Other: standing powered wheelchair evaluation — standing powered wheelchair evaluation

SUMMARY:
The purpose of this study was to explore the experiences of standing powered wheelchair users with spinal cord injury.

DETAILED DESCRIPTION:
There is limited research exploring the comfort, satisfaction, adverse effects, need for repair, and benefit in terms of secondary complications in standing powered wheelchair users with spinal cord injury.

The purpose of this study was to explore the experiences of standing powered wheelchair users with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Post-spinal cord injury period > 1 year

Exclusion Criteria:

- Having cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injury who were prescribed a standing powered wheelchair at a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Wheelchair satisfaction | through study completion, an average of one month
  The patients' level of satisfaction with the features of the standing powered wheelchair will be evaluated with a 5-point Likert scale (from (1) not satisfied at all to (5) very satisfied). Dissatisfaction reason will be noted.
Wheelchair comfort | through study completion, an average of one month
  The patients' overall comfort level while using the standing powered wheelchair and the comfort level in some regions of the body (e.g. back, arms) in the standing position will be evaluated with a 5-point Likert scale (from (1) not satisfied at all to (5) very satisfied).
Wheelchair repair | through study completion, an average of one month
  Participants will be asked whether the standing powered wheelchair needs repairs and the area repaired.
Adverse and positive experiences | through study completion, an average of one month
  Participants will be asked about their adverse and positive experiences with the use of standing powered wheelchair

CONTACTS AND LOCATIONS:
Overall Officials: Merve Örücü Atar, MD, Principal Investigator — Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)